CLINICAL TRIAL: NCT01337596
Title: A Safety, Tolerability, and Pharmacokinetic Study of Single, Escalating Subcutaneous Doses of LY2951742 in Healthy Volunteers
Brief Title: A Study of LY2951742 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14248; I5Q-MC-CGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2012-05

CONDITIONS: Migraines
Keywords: pain; neuropathic pain; headaches
MeSH Terms: conditions — Migraine Disorders; Pain; Neuralgia; Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Single dose 1 milligram (mg) LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose 5 mg LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose 25 mg LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose 75 mg LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose 200 mg LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose 600 mg LY2951742 (Experimental): Administered single subcutaneous injection
  Interventions: Drug: LY2951742
- Single dose placebo (Placebo Comparator): Administered single subcutaneous injection
  Interventions: Drug: Placebo
- Multiple dose placebo (Placebo Comparator): Administered subcutaneously every 2 weeks for 6 weeks (4 doses)
  Interventions: Drug: Placebo
- 150 mg LY2951742 (Experimental): Administered subcutaneously every 2 weeks for 6 weeks (4 doses)
  Interventions: Drug: LY2951742

INTERVENTIONS:
Drug: LY2951742 — Administered subcutaneously
  Arms: 150 mg LY2951742; Single dose 1 milligram (mg) LY2951742; Single dose 200 mg LY2951742; Single dose 25 mg LY2951742; Single dose 5 mg LY2951742; Single dose 600 mg LY2951742; Single dose 75 mg LY2951742
Drug: Placebo — Administered subcutaneously
  Arms: Multiple dose placebo; Single dose placebo

SUMMARY:
To evaluate the safety and tolerability of LY2951742 given as single or multiple subcutaneous injection in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Are healthy Caucasian males, as determined by medical history and physical examination
* Agree to use a reliable method of birth control (e.g. condom AND additional contraception method to be used by respective partner) during the study and for 3 months following the last dose of the investigational product
* Have a body mass index (BMI) greater than 19 kilogram/square meter (kg/m^2)
* Have clinical laboratory test results within normal reference range for the population or investigator site
* Have venous access sufficient to allow for blood sampling
* Are willing to follow study procedures including no drugs (exception of study drug) 72 hours prior to initiation of the laser doppler imaging (LDI) procedure, no chocolate, alcohol or caffeine containing products 12 hours prior to initiation of the laser doppler imaging (LDI) procedure, and complete a 4 hour fast prior to initiation of the laser doppler imaging (LDI) procedure
* Have suitable skin characteristics for the dermal capsaicin challenge and have demonstrated a 100 percent increase in dermal flow following capsaicin challenge as part of the screening procedures and measured by laser doppler imaging (LDI)

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are persons who have previously received the investigational product in this study, have completed or withdrawn from this study investigating LY2951742
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study including QTc greater than 450 milliseconds (msec) (male), history of congenital long QT syndrome or other conduction abnormality
* Have abnormal vital signs as determined by the investigator
* Have a history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders (including migraine) that would constitute a risk when taking the study medication; or of interfering with the interpretation of data study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of:

  1. Human immunodeficiency virus infection and/or positive human immunodeficiency virus (HIV) antibodies
  2. Hepatitis C and/or positive hepatitis C antibody
  3. Hepatitis B and/or positive hepatitis B surface antigen
* Intend to use over-the-counter or prescription medication that may interfere with study safety assessments or other measurements within 7 days prior to dosing and during the study (example: systemic glucocorticoids, immunomodulatory drugs, drugs with propensity for dermal reactions, and drugs with known liver toxicity).
* Have donated blood of more than 500 milliliter (mL) or has undergone major surgery
* The use of caffeine containing products and alcohol is not allowed from 12 hours prior to all study visits and during in clinic stays. All other times, alcohol consumption and caffeine intake are limited to no more than 2 alcoholic beverages or equivalent (beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits (25 milliliter [mL/1 ounce]) per day and caffeinated beverages will be limited to no more than 2 units per day amounts (1 unit=120 milligrams [mg] of caffeine). Strenuous activity is not allowed from 1 week prior to admission until the follow-up visit.
* Are smokers within the previous 6 months
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer)prior to dosing or have received a vaccination within 1 month
* Have a history of multiple or severe allergies or has had an anaphylactic reaction or intolerability to prescription or non-prescription drugs or food
* Are immunocompromised
* Have had cancer or within the past 5 years
* Have a history of significant allergies, in particular to ethanol or sensitivity to the fruits of capsicum plants (example: chili peppers)
* Have eczema, scleroderma, psoriasis, dermatitis, keloids, tumors, ulcers, burns, flaps, or grafts on their forearm or other abnormality of the skin which may interfere with the study assessments
* Cannot avoid excess tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and cannot cover forearms for 24 hours prior to treatment period
* Have excessive hair growth on the volar surface of the forearm or subjects currently using lotions, oils, depilatory preparations, or other topical treatments on a regular basis which cannot be discontinued for the duration of the study; subject has used any topical treatments within 7 days of the start of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg Single Dose LY2951742: Single dose 1 milligram (mg) LY2951742 administered subcutaneously.
- 5 mg Single Dose LY2951742: Single dose 5 mg LY2951742 administered subcutaneously.
- 25 mg Single Dose LY2951742: Single dose 25 mg LY2951742 administered subcutaneously.
- 75 mg Single Dose LY2951742: Single dose 75 mg LY2951742 administered subcutaneously.
- 200 mg Single Dose LY2951742: Single dose 200 mg LY2951742 administered subcutaneously.
- 600 mg Single Dose LY2951742: Single dose 600 mg LY2951742 administered subcutaneously.
- Placebo Single Dose: Single dose matched placebo administered subcutaneously.
- Placebo Multiple Dose: Multiple dose matched placebo administered subcutaneously every 2 weeks for 6 weeks (4 doses).
- 150 mg Multiple Dose LY2951742: Multiple dose 150 mg LY2951742 administered subcutaneously every 2 weeks for 6 weeks (4 doses).
Period: Overall Study
Arm/Group | 1 mg Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742 | Placebo Single Dose | Placebo Multiple Dose | 150 mg Multiple Dose LY2951742
Started | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7
Safety Population | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7
Completed | 7 | 7 | 7 | 7 | 5 | 7 | 12 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 mg Single Dose LY2951742: Single dose 1 mg LY2951742 administered subcutaneously.
- Total: Total of all reporting groups
Arm/Group | 1 mg Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742 | Placebo Single Dose | Placebo Multiple Dose | 150 mg Multiple Dose LY2951742 | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (11.7) | 29.0 (7.5) | 31.9 (14.3) | 30.9 (10.5) | 37.0 (14.6) | 33.9 (13.9) | 30.8 (10.0) | 22.5 (0.7) | 22.4 (1.6) | 30.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7 | 63
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and other non-serious adverse events (AEs). A summary of serious and all other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: Baseline up to 6 months (study completion)
Population: Safety Population: All participants who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Groups:
- 1 Milligram (mg) Single Dose LY2951742: Single dose 1 mg LY2951742 administered subcutaneously.
Arm/Group | 1 Milligram (mg) Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742 | Placebo Single Dose | Placebo Multiple Dose | 150 mg Multiple Dose LY2951742
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 2 | 7
participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other Non-Serious Adverse Events | 6 | 5 | 7 | 4 | 7 | 5 | 9 | 2 | 7

2. Secondary Outcome: Single Dose Pharmacokinetics of LY2951742 Maximal Concentration (Cmax)
Time Frame: Day 1 up to Day 84 or early discontinuation
Population: Pharmacokinetic (PK) Population: All participants who received single dose LY2951742 study drug with interpretable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 75 mg Single Dose LY2951742: Single dose 175mg LY2951742 administered subcutaneously.
Arm/Group | 1 mg Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
nanogram per milliliter (ng/mL) | 95.60 (21.26) | 404.61 (34.45) | 1995.35 (44.48) | 5920.79 (48.51) | 13750.14 (40.72) | 45039.42 (22.52)

3. Secondary Outcome: Single Dose Pharmacokinetics of LY2951742 Area Under the Curve (AUC)
Time Frame: Day 1 up to Day 84 or early discontinuation
Population: PK Population: All participants who received single dose LY2951742 study drug with interpretable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*day per milliliter (ng*day/mL)
Arm/Group | 1 mg Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
nanogram*day per milliliter (ng*day/mL) | 4718.4 (11.6) | 19743.5 (29.7) | 92310.1 (32.7) | 263144.2 (44.7) | 624419.4 (39.8) | 2280259.7 (9.8)

4. Secondary Outcome: Multiple Dose Pharmacokinetics of LY2951742 Maximal Concentration (Cmax)
Time Frame: Day 43 up to Day 57
Population: PK Population: All participants who received multiple doses LY2951742 study drug with interpretable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150 mg Multiple Dose LY2951742
Number analyzed (Participants) | 7
ng/mL | 36846.420 (14.878)

5. Secondary Outcome: Multiple Dose Pharmacokinetics of LY2951742 Area Under the Curve (AUC)
Time Frame: Day 43 up to Day 57
Population: PK Population: All participants who received multiple dose LY2951742 study drug with interpretable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*day/mL
Arm/Group | 150 mg Multiple Dose LY2951742
Number analyzed (Participants) | 7
ng*day/mL | 1806501.8 (20.4)

ADVERSE EVENTS:
Arm/Group | 1 mg Single Dose LY2951742 | 5 mg Single Dose LY2951742 | 25 mg Single Dose LY2951742 | 75 mg Single Dose LY2951742 | 200 mg Single Dose LY2951742 | 600 mg Single Dose LY2951742 | Placebo Single Dose | Placebo Multiple Dose | 150 mg Multiple Dose LY2951742
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/12 | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 5/7 | 7/7 | 4/7 | 7/7 | 5/7 | 9/12 | 2/2 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Single Dose LY2951742 (N=7) | 5 mg Single Dose LY2951742 (N=7) | 25 mg Single Dose LY2951742 (N=7) | 75 mg Single Dose LY2951742 (N=7) | 200 mg Single Dose LY2951742 (N=7) | 600 mg Single Dose LY2951742 (N=7) | Placebo Single Dose (N=12) | Placebo Multiple Dose (N=2) | 150 mg Multiple Dose LY2951742 (N=7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin e increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 4 (4) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days